CLINICAL TRIAL: NCT04496102
Title: Comparison of Efficacy Between Cemented and Cementless Total Knee Arthroplasty in Bilateral Total Knee Arthroplasty. A Prospective Randomized Controlled Trial
Brief Title: Cemented vs Cementless in Bilateral TKA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Thammasat University (Other)
Responsible Party: Principal Investigator, Supakit Kanitnate, Principal Investigator, Thammasat University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OrthoTU12
Record Dates: First submitted 2020-07-17; First posted 2020-08-03 (Actual); Last update posted 2020-08-03 (Actual); Status verified 2020-07

CONDITIONS: Osteoarthritis; Total Knee Arthroplasty
Keywords: cemented; cementless; total knee arthroplasty; short term outcome; functional outcome
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Cemented TKA (Active Comparator): Cemented TKA (Triathlon, Stryker) include patellar resurfacing
  Interventions: Device: Triathlon
- Cementless TKA (Experimental): Cementless TKA (Triathlon Tritanium, Stryker) include patellar resurfacing
  Interventions: Device: Triathlon

INTERVENTIONS:
Device: Triathlon — Modern TKA design (Triathlon) with patellar resurfacing

SUMMARY:
To compare the functional outcomes between cemented and cementless TKA in bilateral knee replacement patient.

DETAILED DESCRIPTION:
To compare early functional outcomes, radiographic finding and operative time between cemented and cementless modern implant in sequential bilateral total kee arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* ASA status 1 or 2
* Diagnosed with bilateral osteoarthritis of the knees
* Participant understand and consent to the protocol of the trial

Exclusion Criteria:

* Morbid obesity (BMI >40)
* Inflammatory arthritis
* Osteoporosis
* Metabolic bone disease
* Bone defect that seen from radiographs

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Compare mean Forgotten joint score between 2 groups | at 1 year
  The total score ranges from 0-100, where a high score is the best outcome

SECONDARY OUTCOMES:
Operative time | intra-operative assessment
modified the Western Ontario and McMaster Universities Osteoarthritis Index score | post-op 2, 6 week, 3, 6, 12 month
  The total score ranges from 0-96, where a high score is the worse outcome
Pain level | Once daily 1-14 days after surgery then once a week until 3 months
  VAS for pain (0-100)
Range of knee motion | post-op 2, 6 week, 3, 6, 12 month
  flexion and extension (degrees) which measured by long goniometer
complication | until 1 year after surgery
  such as fracture, infection, stiffness
Radiological finding | post-op 2, 6 week, 3, 6, 12 month
  Radiolucent line at femoral, tibial and patellar components which measured from radiolucent intervals (measured in millimetres) between the cement or prostheses and the bone according to the knee society total knee arthroplasty roentgenographic evaluation and scoring system

CONTACTS AND LOCATIONS:
Locations (1):
- Thammasat University, Khlong Luang, Changwat Pathum Thani, Thailand

IPD SHARING:
Plan to Share IPD: No